CLINICAL TRIAL: NCT01302210
Title: Detection, Education, Research and Decolonization Without Isolation in Long-term Care to Control(DERAIL)MRSA
Brief Title: Detection, Education, Research and Decolonization Without Isolation in Long-term Care Facilities
Acronym: DERAIL_MRSA
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: AHRQ 1R18HSO19968-01
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Methicillin Resistant Staphylococcus Aureus
Keywords: MRSA; Cluster Randomized Trial; Infection Control Intervention
MeSH Terms: interventions — Mupirocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention: Active surveillance testing for MRSA and decolonization of positive subjects
  Interventions: Drug: Decolonization
- control: Usual standard of care

INTERVENTIONS:
Drug: Decolonization — 5 day regimen of mupirocin calcium 2% twice daily to the nares and any open wound plus bath or shower with 4% chlorhexidine used as a liquid soap
  Other Names: Mupirocin
  Groups: Intervention

SUMMARY:
Our hypothesis for the DERAIL MRSA program is that one can safely remove the colonization risk from nearly all residents (patients) in a way that does not interfere with the desired life-style for persons in these facilities and thereby reduce the risk of infection and lower the cost of care by avoiding preventable disease.

DETAILED DESCRIPTION:
The primary endpoint will be measuring the reduction in MRSA colonization prevalence (percentage rate) in the intervention arm as compared to the control arm. One secondary endpoint is to compare the rate of MRSA disease (number of infections per 1,000 patients and 10,000 patient days) in the intervention and control arms. The other secondary endpoint is to determine the cost of MRSA screening and decolonization and compare it to the cost of MRSA disease treatment (both medication cost and the expense of any needed hospitalization for therapy of MRSA infection therapy) in the control arm. Achieving our primary goal of MRSA control will also demonstrate two secondary goals wthe investigators aim to achieve: one being that a scientific, planned approach to the issue of specific healthcare-associated infection in LTCFs can resolve these problems and the other that a partnership between acute and long-term care (e.g., ongoing relationship spanning at least 5 years) is beneficial in dealing with patient safety and quality practices across the United Sates Healthcare continuum.

ELIGIBILITY:
Inclusion Criteria:

* All patients in 18 LTCF nursing units randomly selected as intervention or control units

Exclusion Criteria:

* Patients that choose not to be included in the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22302 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
To record the effectiveness of an admission testing and immediate decolonization of positive persons protocol for reducing MRSA colonization prevalence in long term care facilities (LTCF's) | 12 months and 24 months
  Infection Control cluster randomized trial: measuring the reduction in MRSA colonization prevalence (rate) in the intervention arm as compared to the control arm

SECONDARY OUTCOMES:
To further develop an Infection Control Outreach Program designed to provide expert guidance on infectious disease prevention specific to LTCF's | 2 years
  Compare the rate of MRSA disease in the intervention and control arms. Determine the cost of MRSA screening and decolonization and compare it to the cost of MRSA disease treatment (both medication cost and the expense of any needed hospitalization for therapy of MRSA infection therapy) in the control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Lance R Peterson, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem Research Institute, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capitano B, Leshem OA, Nightingale CH, Nicolau DP. Cost effect of managing methicillin-resistant Staphylococcus aureus in a long-term care facility. J Am Geriatr Soc. 2003 Jan;51(1):10-6. doi: 10.1034/j.1601-5215.2002.51003.x. PMID 12534839
- [Background] Kauffman CA, Terpenning MS, He X, Zarins LT, Ramsey MA, Jorgensen KA, Sottile WS, Bradley SF. Attempts to eradicate methicillin-resistant Staphylococcus aureus from a long-term-care facility with the use of mupirocin ointment. Am J Med. 1993 Apr;94(4):371-8. doi: 10.1016/0002-9343(93)90147-h. PMID 8475930
- [Background] Vriens M, Blok H, Fluit A, Troelstra A, Van Der Werken C, Verhoef J. Costs associated with a strict policy to eradicate methicillin-resistant Staphylococcus aureus in a Dutch University Medical Center: a 10-year survey. Eur J Clin Microbiol Infect Dis. 2002 Nov;21(11):782-6. doi: 10.1007/s10096-002-0811-4. Epub 2002 Nov 8. PMID 12461587
- [Background] Smith PW, Bennett G, Bradley S, Drinka P, Lautenbach E, Marx J, Mody L, Nicolle L, Stevenson K; SHEA; APIC. SHEA/APIC guideline: infection prevention and control in the long-term care facility, July 2008. Infect Control Hosp Epidemiol. 2008 Sep;29(9):785-814. doi: 10.1086/592416. No abstract available. PMID 18767983
- [Background] Siegel JD, Rhinehart E, Jackson M, Chiarello L; Health Care Infection Control Practices Advisory Committee. 2007 Guideline for Isolation Precautions: Preventing Transmission of Infectious Agents in Health Care Settings. Am J Infect Control. 2007 Dec;35(10 Suppl 2):S65-164. doi: 10.1016/j.ajic.2007.10.007. No abstract available. PMID 18068815
- [Background] Haley RW, Culver DH, White JW, Morgan WM, Emori TG. The nationwide nosocomial infection rate. A new need for vital statistics. Am J Epidemiol. 1985 Feb;121(2):159-67. doi: 10.1093/oxfordjournals.aje.a113988. PMID 4014113
- [Background] Strausbaugh LJ, Joseph CL. The burden of infection in long-term care. Infect Control Hosp Epidemiol. 2000 Oct;21(10):674-9. doi: 10.1086/501712. PMID 11083186
- [Background] Haley RW, Culver DH, White JW, Morgan WM, Emori TG, Munn VP, Hooton TM. The efficacy of infection surveillance and control programs in preventing nosocomial infections in US hospitals. Am J Epidemiol. 1985 Feb;121(2):182-205. doi: 10.1093/oxfordjournals.aje.a113990. PMID 4014115
- [Background] John JF Jr, Ribner BS. Antibiotic resistance in long-term care facilities. Infect Control Hosp Epidemiol. 1991 Apr;12(4):245-50. doi: 10.1086/646332. No abstract available. PMID 1905739
- [Background] Muder RR, Brennen C, Wagener MM, Vickers RM, Rihs JD, Hancock GA, Yee YC, Miller JM, Yu VL. Methicillin-resistant staphylococcal colonization and infection in a long-term care facility. Ann Intern Med. 1991 Jan 15;114(2):107-12. doi: 10.7326/0003-4819-114-2-1-107. PMID 1984384
- [Background] Bradley SF, Terpenning MS, Ramsey MA, Zarins LT, Jorgensen KA, Sottile WS, Schaberg DR, Kauffman CA. Methicillin-resistant Staphylococcus aureus: colonization and infection in a long-term care facility. Ann Intern Med. 1991 Sep 15;115(6):417-22. doi: 10.7326/0003-4819-115-6-417. PMID 1908198
- [Background] Strausbaugh LJ, Jacobson C, Sewell DL, Potter S, Ward TT. Methicillin-resistant Staphylococcus aureus in extended-care facilities: experiences in a Veterans' Affairs nursing home and a review of the literature. Infect Control Hosp Epidemiol. 1991 Jan;12(1):36-45. doi: 10.1086/646236. PMID 1999642
- [Background] Boyce JM. Methicillin-resistant Staphylococcus aureus in hospitals and long-term care facilities: microbiology, epidemiology, and preventive measures. Infect Control Hosp Epidemiol. 1992 Dec;13(12):725-37. doi: 10.1086/648346. No abstract available. PMID 1289400
- [Background] Trick WE, Weinstein RA, DeMarais PL, Kuehnert MJ, Tomaska W, Nathan C, Rice TW, McAllister SK, Carson LA, Jarvis WR. Colonization of skilled-care facility residents with antimicrobial-resistant pathogens. J Am Geriatr Soc. 2001 Mar;49(3):270-6. doi: 10.1046/j.1532-5415.2001.4930270.x. PMID 11300237
- [Background] Stone ND, Lewis DR, Lowery HK, Darrow LA, Kroll CM, Gaynes RP, Jernigan JA, McGowan JE Jr, Tenover FC, Richards CL Jr. Importance of bacterial burden among methicillin-resistant Staphylococcus aureus carriers in a long-term care facility. Infect Control Hosp Epidemiol. 2008 Feb;29(2):143-8. doi: 10.1086/526437. PMID 18179369
- [Background] Brugnaro P, Fedeli U, Pellizzer G, Buonfrate D, Rassu M, Boldrin C, Parisi SG, Grossato A, Palu G, Spolaore P. Clustering and risk factors of methicillin-resistant Staphylococcus aureus carriage in two Italian long-term care facilities. Infection. 2009 Jun;37(3):216-21. doi: 10.1007/s15010-008-8165-1. Epub 2008 Dec 9. PMID 19148574
- [Background] March A, Aschbacher R, Dhanji H, Livermore DM, Bottcher A, Sleghel F, Maggi S, Noale M, Larcher C, Woodford N. Colonization of residents and staff of a long-term-care facility and adjacent acute-care hospital geriatric unit by multiresistant bacteria. Clin Microbiol Infect. 2010 Jul;16(7):934-44. doi: 10.1111/j.1469-0691.2009.03024.x. Epub 2009 Aug 17. PMID 19686277
- [Background] Suetens C, Niclaes L, Jans B, Verhaegen J, Schuermans A, Van Eldere J, Buntinx F. Methicillin-resistant Staphylococcus aureus colonization is associated with higher mortality in nursing home residents with impaired cognitive status. J Am Geriatr Soc. 2006 Dec;54(12):1854-60. doi: 10.1111/j.1532-5415.2006.00972.x. PMID 17198490
- [Background] Capitano B, Nicolau DP. Evolving epidemiology and cost of resistance to antimicrobial agents in long-term care facilities. J Am Med Dir Assoc. 2003 May-Jun;4(3 Suppl):S90-9. doi: 10.1097/01.JAM.0000066029.00660.5A. No abstract available. PMID 12854980
- [Background] Hughes CM, Smith MB, Tunney MM. Infection control strategies for preventing the transmission of meticillin-resistant Staphylococcus aureus (MRSA) in nursing homes for older people. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD006354. doi: 10.1002/14651858.CD006354.pub2. PMID 18254100
- [Background] Gorwitz RJ, Kruszon-Moran D, McAllister SK, McQuillan G, McDougal LK, Fosheim GE, Jensen BJ, Killgore G, Tenover FC, Kuehnert MJ. Changes in the prevalence of nasal colonization with Staphylococcus aureus in the United States, 2001-2004. J Infect Dis. 2008 May 1;197(9):1226-34. doi: 10.1086/533494. PMID 18422434
- [Background] Davis KA, Stewart JJ, Crouch HK, Florez CE, Hospenthal DR. Methicillin-resistant Staphylococcus aureus (MRSA) nares colonization at hospital admission and its effect on subsequent MRSA infection. Clin Infect Dis. 2004 Sep 15;39(6):776-82. doi: 10.1086/422997. Epub 2004 Aug 27. PMID 15472807
- [Background] Huang SS, Platt R. Risk of methicillin-resistant Staphylococcus aureus infection after previous infection or colonization. Clin Infect Dis. 2003 Feb 1;36(3):281-5. doi: 10.1086/345955. Epub 2003 Jan 17. PMID 12539068
- [Background] Datta R, Huang SS. Risk of infection and death due to methicillin-resistant Staphylococcus aureus in long-term carriers. Clin Infect Dis. 2008 Jul 15;47(2):176-81. doi: 10.1086/589241. PMID 18532892
- [Background] Cosgrove SE, Sakoulas G, Perencevich EN, Schwaber MJ, Karchmer AW, Carmeli Y. Comparison of mortality associated with methicillin-resistant and methicillin-susceptible Staphylococcus aureus bacteremia: a meta-analysis. Clin Infect Dis. 2003 Jan 1;36(1):53-9. doi: 10.1086/345476. Epub 2002 Dec 13. PMID 12491202
- [Background] Ben-David D, Novikov I, Mermel LA. Are there differences in hospital cost between patients with nosocomial methicillin-resistant Staphylococcus aureus bloodstream infection and those with methicillin-susceptible S. aureus bloodstream infection? Infect Control Hosp Epidemiol. 2009 May;30(5):453-60. doi: 10.1086/596731. PMID 19344266
- [Background] Klevens RM, Morrison MA, Nadle J, Petit S, Gershman K, Ray S, Harrison LH, Lynfield R, Dumyati G, Townes JM, Craig AS, Zell ER, Fosheim GE, McDougal LK, Carey RB, Fridkin SK; Active Bacterial Core surveillance (ABCs) MRSA Investigators. Invasive methicillin-resistant Staphylococcus aureus infections in the United States. JAMA. 2007 Oct 17;298(15):1763-71. doi: 10.1001/jama.298.15.1763. PMID 17940231
- [Background] Kaye KS, Anderson DJ, Choi Y, Link K, Thacker P, Sexton DJ. The deadly toll of invasive methicillin-resistant Staphylococcus aureus infection in community hospitals. Clin Infect Dis. 2008 May 15;46(10):1568-77. doi: 10.1086/587673. PMID 18419491
- [Background] Humphreys H, Grundmann H, Skov R, Lucet JC, Cauda R. Prevention and control of methicillin-resistant Staphylococcus aureus. Clin Microbiol Infect. 2009 Feb;15(2):120-4. doi: 10.1111/j.1469-0691.2009.02699.x. PMID 19291143
- [Background] Delorme T, Rose S, Senita J, Callahan C, Nasr P. Epidemiology and susceptibilities of methicillin-resistant Staphylococcus aureus in Northeastern Ohio. Am J Clin Pathol. 2009 Nov;132(5):668-77. doi: 10.1309/AJCPQ46ZPQXVHHNC. PMID 19846806
- [Background] Lindsay JA. Genomic variation and evolution of Staphylococcus aureus. Int J Med Microbiol. 2010 Feb;300(2-3):98-103. doi: 10.1016/j.ijmm.2009.08.013. Epub 2009 Oct 7. PMID 19811948
- [Background] Sung JM, Lloyd DH, Lindsay JA. Staphylococcus aureus host specificity: comparative genomics of human versus animal isolates by multi-strain microarray. Microbiology (Reading). 2008 Jul;154(Pt 7):1949-1959. doi: 10.1099/mic.0.2007/015289-0. PMID 18599823
- [Background] Grundmann H, Aanensen DM, van den Wijngaard CC, Spratt BG, Harmsen D, Friedrich AW; European Staphylococcal Reference Laboratory Working Group. Geographic distribution of Staphylococcus aureus causing invasive infections in Europe: a molecular-epidemiological analysis. PLoS Med. 2010 Jan 12;7(1):e1000215. doi: 10.1371/journal.pmed.1000215. PMID 20084094
- [Background] Deurenberg RH, Vink C, Kalenic S, Friedrich AW, Bruggeman CA, Stobberingh EE. The molecular evolution of methicillin-resistant Staphylococcus aureus. Clin Microbiol Infect. 2007 Mar;13(3):222-35. doi: 10.1111/j.1469-0691.2006.01573.x. PMID 17391376
- [Background] Feil EJ, Cooper JE, Grundmann H, Robinson DA, Enright MC, Berendt T, Peacock SJ, Smith JM, Murphy M, Spratt BG, Moore CE, Day NP. How clonal is Staphylococcus aureus? J Bacteriol. 2003 Jun;185(11):3307-16. doi: 10.1128/JB.185.11.3307-3316.2003. PMID 12754228
- [Background] Feil EJ. Small change: keeping pace with microevolution. Nat Rev Microbiol. 2004 Jun;2(6):483-95. doi: 10.1038/nrmicro904. No abstract available. PMID 15152204
- [Background] Robicsek A, Beaumont JL, Thomson RB Jr, Govindarajan G, Peterson LR. Topical therapy for methicillin-resistant Staphylococcus aureus colonization: impact on infection risk. Infect Control Hosp Epidemiol. 2009 Jul;30(7):623-32. doi: 10.1086/597550. PMID 19496730
- [Background] Peterson LR, Hacek DM, Robicsek A. 5 Million Lives Campaign. Case study: an MRSA intervention at Evanston Northwestern Healthcare. Jt Comm J Qual Patient Saf. 2007 Dec;33(12):732-8. doi: 10.1016/s1553-7250(07)33088-2. PMID 18200898
- [Background] Chang S, Sethi AK, Eckstein BC, Stiefel U, Cadnum JL, Donskey CJ. Skin and environmental contamination with methicillin-resistant Staphylococcus aureus among carriers identified clinically versus through active surveillance. Clin Infect Dis. 2009 May 15;48(10):1423-8. doi: 10.1086/598505. PMID 19364286
- [Background] Smith NH, Gordon SV, de la Rua-Domenech R, Clifton-Hadley RS, Hewinson RG. Bottlenecks and broomsticks: the molecular evolution of Mycobacterium bovis. Nat Rev Microbiol. 2006 Sep;4(9):670-81. doi: 10.1038/nrmicro1472. PMID 16912712
- [Background] Bowler WA, Bresnahan J, Bradfish A, Fernandez C. An integrated approach to methicillin-resistant Staphylococcus aureus control in a rural, regional-referral healthcare setting. Infect Control Hosp Epidemiol. 2010 Mar;31(3):269-75. doi: 10.1086/650445. PMID 20102280
- [Background] Robicsek A, Beaumont JL, Paule SM, Hacek DM, Thomson RB Jr, Kaul KL, King P, Peterson LR. Universal surveillance for methicillin-resistant Staphylococcus aureus in 3 affiliated hospitals. Ann Intern Med. 2008 Mar 18;148(6):409-18. doi: 10.7326/0003-4819-148-6-200803180-00003. PMID 18347349
- [Background] Peterson LR, Diekema DJ. To screen or not to screen for methicillin-resistant Staphylococcus aureus. J Clin Microbiol. 2010 Mar;48(3):683-9. doi: 10.1128/JCM.02516-09. Epub 2010 Jan 13. PMID 20071548
- [Background] Bocher S, Skov RL, Knudsen MA, Guardabassi L, Molbak K, Schouenborg P, Sorum M, Westh H. The search and destroy strategy prevents spread and long-term carriage of methicillin-resistant Staphylococcus aureus: results from the follow-up screening of a large ST22 (E-MRSA 15) outbreak in Denmark. Clin Microbiol Infect. 2010 Sep;16(9):1427-34. doi: 10.1111/j.1469-0691.2009.03137.x. PMID 20041904
- [Background] Jernigan JA, Titus MG, Groschel DH, Getchell-White S, Farr BM. Effectiveness of contact isolation during a hospital outbreak of methicillin-resistant Staphylococcus aureus. Am J Epidemiol. 1996 Mar 1;143(5):496-504. doi: 10.1093/oxfordjournals.aje.a008770. PMID 8610665
- [Background] Stosor V, Kruszynski J, Suriano T, Noskin GA, Peterson LR. Molecular epidemiology of vancomycin-resistant enterococci: a 2-year perspective. Infect Control Hosp Epidemiol. 1999 Oct;20(10):653-9. doi: 10.1086/501560. PMID 10530641
- [Background] Savor C, Pfaller MA, Kruszynski JA, Hollis RJ, Noskin GA, Peterson LR. Comparison of genomic methods for differentiating strains of Enterococcus faecium: assessment using clinical epidemiologic data. J Clin Microbiol. 1998 Nov;36(11):3327-31. doi: 10.1128/JCM.36.11.3327-3331.1998. PMID 9774587
- [Background] Jaggi P, Paule SM, Peterson LR, Tan TQ. Characteristics of Staphylococcus aureus infections, Chicago Pediatric Hospital. Emerg Infect Dis. 2007 Feb;13(2):311-4. doi: 10.3201/eid1302.060295. PMID 17479900
- [Background] Hubbard AE, Ahern J, Fleischer NL, Van der Laan M, Lippman SA, Jewell N, Bruckner T, Satariano WA. To GEE or not to GEE: comparing population average and mixed models for estimating the associations between neighborhood risk factors and health. Epidemiology. 2010 Jul;21(4):467-74. doi: 10.1097/EDE.0b013e3181caeb90. PMID 20220526
- [Background] Roy J, Lin X, Ryan LM. Scaled marginal models for multiple continuous outcomes. Biostatistics. 2003 Jul;4(3):371-83. doi: 10.1093/biostatistics/4.3.371. PMID 12925505
- [Background] Paule SM, Mehta M, Hacek DM, Gonzalzles TM, Robicsek A, Peterson LR. Chromogenic media vs real-time PCR for nasal surveillance of methicillin-resistant Staphylococcus aureus: impact on detection of MRSA-positive persons. Am J Clin Pathol. 2009 Apr;131(4):532-9. doi: 10.1309/AJCP18ONZUTDUGAQ. PMID 19289589
- [Background] Mody L, Kauffman CA, McNeil SA, Galecki AT, Bradley SF. Mupirocin-based decolonization of Staphylococcus aureus carriers in residents of 2 long-term care facilities: a randomized, double-blind, placebo-controlled trial. Clin Infect Dis. 2003 Dec 1;37(11):1467-74. doi: 10.1086/379325. Epub 2003 Nov 6. PMID 14614669
- [Background] Suetens C, Niclaes L, Jans B, Verhaegen J, Schuermans A, Van Eldere J, Vandenbroucke JP, Buntinx F. Determinants of methicillin-resistant Staphylococcus aureus carriage in nursing homes. Age Ageing. 2007 May;36(3):327-30. doi: 10.1093/ageing/afm013. Epub 2007 Mar 29. No abstract available. PMID 17395619
- [Background] Robicsek A, Suseno M, Beaumont JL, Thomson RB Jr, Peterson LR. Prediction of methicillin-resistant Staphylococcus aureus involvement in disease sites by concomitant nasal sampling. J Clin Microbiol. 2008 Feb;46(2):588-92. doi: 10.1128/JCM.01746-07. Epub 2007 Dec 5. PMID 18057132
- [Background] Baker SE, Brecher SM, Robillard E, Strymish J, Lawler E, Gupta K. Extranasal methicillin-resistant Staphylococcus aureus colonization at admission to an acute care Veterans Affairs hospital. Infect Control Hosp Epidemiol. 2010 Jan;31(1):42-6. doi: 10.1086/649222. PMID 19954335
- [Background] Miller MA, Dascal A, Portnoy J, Mendelson J. Development of mupirocin resistance among methicillin-resistant Staphylococcus aureus after widespread use of nasal mupirocin ointment. Infect Control Hosp Epidemiol. 1996 Dec;17(12):811-3. doi: 10.1086/647242. PMID 8985769
- [Background] McConeghy KW, Mikolich DJ, LaPlante KL. Agents for the decolonization of methicillin-resistant Staphylococcus aureus. Pharmacotherapy. 2009 Mar;29(3):263-80. doi: 10.1592/phco.29.3.263. PMID 19249946
- [Background] Urth T, Juul G, Skov R, Schonheyder HC. Spread of a methicillin-resistant Staphylococcus aureus ST80-IV clone in a Danish community. Infect Control Hosp Epidemiol. 2005 Feb;26(2):144-9. doi: 10.1086/502518. PMID 15756884
- [Background] Boelaert JR. Staphylococcus aureus infection in haemodialysis patients. Mupirocin as a topical strategy against nasal carriage: a review. J Chemother. 1994 Apr;6 Suppl 2:19-24. PMID 7799051
- [Background] Bode LG, Kluytmans JA, Wertheim HF, Bogaers D, Vandenbroucke-Grauls CM, Roosendaal R, Troelstra A, Box AT, Voss A, van der Tweel I, van Belkum A, Verbrugh HA, Vos MC. Preventing surgical-site infections in nasal carriers of Staphylococcus aureus. N Engl J Med. 2010 Jan 7;362(1):9-17. doi: 10.1056/NEJMoa0808939. PMID 20054045
- [Background] Hacek DM, Robb WJ, Paule SM, Kudrna JC, Stamos VP, Peterson LR. Staphylococcus aureus nasal decolonization in joint replacement surgery reduces infection. Clin Orthop Relat Res. 2008 Jun;466(6):1349-55. doi: 10.1007/s11999-008-0210-y. Epub 2008 Mar 18. PMID 18347889
- [Background] Ridenour G, Lampen R, Federspiel J, Kritchevsky S, Wong E, Climo M. Selective use of intranasal mupirocin and chlorhexidine bathing and the incidence of methicillin-resistant Staphylococcus aureus colonization and infection among intensive care unit patients. Infect Control Hosp Epidemiol. 2007 Oct;28(10):1155-61. doi: 10.1086/520102. Epub 2007 Aug 1. PMID 17828692
- [Background] Eveillard M, Charru P, Rufat P, Hippeaux MC, Lancien E, Benselama F, Branger C. Methicillin-resistant Staphylococcus aureus carriage in a long-term care facility: hypothesis about selection and transmission. Age Ageing. 2008 May;37(3):294-9. doi: 10.1093/ageing/afn021. Epub 2008 Feb 12. PMID 18270245
- [Background] Munoz-Price LS, Hayden MK, Lolans K, Won S, Calvert K, Lin M, Stemer A, Weinstein RA. Successful control of an outbreak of Klebsiella pneumoniae carbapenemase-producing K. pneumoniae at a long-term acute care hospital. Infect Control Hosp Epidemiol. 2010 Apr;31(4):341-7. doi: 10.1086/651097. PMID 20175685
- [Background] Centers for Disease Control and Prevention (CDC). Trends in tuberculosis--United States, 2004. MMWR Morb Mortal Wkly Rep. 2005 Mar 18;54(10):245-9. PMID 15772584
- [Background] O'Dowd A. NHS may miss target on reducing MRSA by 2008, minister says. BMJ 2006;333(7575:938
- [Background] Peterson LR, Hacek DM, Beaumont JL, Boehm S, Gonzolzaes T-M, Gocht N, Robicsek A. Impact of a 4-Year Universal Surveillance and Decolonization Program to Control Methicillin-Resistant Staphylococcus aureus (MRSA). In Program and Abstracts, Fifth Decennial International Conference on Healthcare-Associated Infection. Atlanta, GA. March 18-22, 2010
- [Background] Perl TM, Cullen JJ, Wenzel RP, Zimmerman MB, Pfaller MA, Sheppard D, Twombley J, French PP, Herwaldt LA; Mupirocin And The Risk Of Staphylococcus Aureus Study Team. Intranasal mupirocin to prevent postoperative Staphylococcus aureus infections. N Engl J Med. 2002 Jun 13;346(24):1871-7. doi: 10.1056/NEJMoa003069. PMID 12063371
- [Background] Robicsek A, Paule SM, Hacek DM, Gonzalzles TM, Thomson RB, Peterson LR. How long after colonization does MRSA disease occur? IN: Program and Abstracts, Forty-eighth Interscience Conference on Antimicrobial Agents and Chemotherapy, Washinton, D.C., October 25-28, 2008. Abstract K-1708.
- [Background] Robicsek A, Hacek DM, Fisher A, Peterson LR. Progression to MRSA infection in asymptomatic carriers (AC) detected through a hospital-based universal surveillance and decolonization program. IN: Program and Abstracts. Forty-fourth Annual Meeting, Infectious Diseases Society of America, Toronto, Canada, October 12-15, 2006. Abstract 390.
- [Background] Hacek D, Paule S, Small M, Gottschall R, Thomson R, Peterson L. Comparison of colisitin naladixic agar (CNA), mannitol salt agar (MS) and phenol mannitol broth with antibiotics (PMB) for the recovery of Staphylococcus aureus (SA) from nasal swabs. Abstracts of the One-hundreth and third Annual Meeting of the American Society for Microbiology,Washinto, DC. May 18-22,2003. Abstract C-323.
- [Background] Paule S, Robicsek A, Suseno M, Kaul KL, Peterson LR. Incidence of mupirocin resistance in methicillin-resistant Staphylococcus aureus (MRSA) during universal surveillance and decolonization. IN: Program and Abstracts, Forty-sixth Interscience Conference on Antimicrobial Agents and Chemotherapy, San Francisco, CA, September 27-30,2006. Abstract C2-1149.
- [Result] Peterson LR, Boehm S, Beaumont JL, Patel PA, Schora DM, Peterson KE, Burdsall D, Hines C, Fausone M, Robicsek A, Smith BA. Reduction of methicillin-resistant Staphylococcus aureus infection in long-term care is possible while maintaining patient socialization: A prospective randomized clinical trial. Am J Infect Control. 2016 Dec 1;44(12):1622-1627. doi: 10.1016/j.ajic.2016.04.251. Epub 2016 Aug 1. PMID 27492790
- [Result] Schora DM, Boehm S, Das S, Patel PA, O'Brien J, Hines C, Burdsall D, Beaumont J, Peterson K, Fausone M, Peterson LR. Impact of Detection, Education, Research and Decolonization without Isolation in Long-term care (DERAIL) on methicillin-resistant Staphylococcus aureus colonization and transmission at 3 long-term care facilities. Am J Infect Control. 2014 Oct;42(10 Suppl):S269-73. doi: 10.1016/j.ajic.2014.05.011. PMID 25239721
- [Result] Das S, Anderson CJ, Grayes A, Mendoza K, Harazin M, Schora DM, Peterson LR. Nasal Carriage of Epidemic Methicillin-Resistant Staphylococcus aureus 15 (EMRSA-15) Clone Observed in Three Chicago-Area Long-Term Care Facilities. Antimicrob Agents Chemother. 2013 Sep;57(9):4551-4553. doi: 10.1128/AAC.00528-13. Epub 2013 Jun 24. PMID 23796939
- See also: Last assessed March 21, 2010 — http://www.idph.state.il.us/healthca/nursinghometestjava.htm
- See also: World Health Organization. The Stop TB strategy. WHO 2006. Last accessed March 13,2010 — http://whqlibdoc.who.int/hq/2006/WHO_HTM_STB_2006.368_eng.pdf